CLINICAL TRIAL: NCT05616312
Title: Validating a "Teach-back" Protocol to Improve Recall in Orthopedic Trauma Patients
Brief Title: Patient Recall After Orthopedic Trauma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, John Sontich, Physician, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY20220951
Record Dates: First submitted 2022-11-07; First posted 2022-11-15 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Education After Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postoperative teach-back educational program (Experimental): Patients will receive teach-back education while they fill out questionnaires.
  Interventions: Behavioral: Educational Teach Back
- Control (No Intervention): Patients will not receive any teach-back education while filling out questionnaires.

INTERVENTIONS:
Behavioral: Educational Teach Back — Patients will receive teach-back education while they fill out questionnaires.
  Arms: Postoperative teach-back educational program

SUMMARY:
The purpose of this study is to evaluate whether receiving education after trauma surgeries affects three things: 1) knowledge about injury and treatment ("recall"), 2) how well patients follow treatment recommendations, and 3) how satisfied patients are with their care. To do so, some participants in this study will receive education, and some will not.

ELIGIBILITY:
Inclusion Criteria:

* Isolated open or closed fracture of the pelvis and/or lower extremity treated surgically

Exclusion Criteria:

* Patient receiving orthopedic care or follow-up at another institution
* Non-English speaking
* Incarcerated (or likely impending incarceration)
* Currently enrolled in a study that does not permit co-enrollment
* Traumatic brain injury, dementia, or other cognitive impairment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2022-10-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of correct answers to the recall-assessing items on the follow-up questionnaire. | Up to 45 minutes
Adherence rate to postoperative weightbearing instructions as measured by patient report. | Up to 180 days post op
Adherence rate to DVT prophylaxis instructions as measured by patient report. | Up to 180 days post op
Mean satisfaction as measured by follow-up questionnaire. | Up to 180 days post op
  Satisfaction will be measured on a Likert scale from 1-5 with 1 being very dissatisfied and 5 being very satisfied with care

CONTACTS AND LOCATIONS:
Overall Officials: John Sontich, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No